CLINICAL TRIAL: NCT01562548
Title: A Proof of Principle Study to Explore the Utility of Guaifenesin in Upper Back Pain
Brief Title: Exploratory Efficacy Study of Guaifenesin in Upper Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: A3940666
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-03

CONDITIONS: Upper Back Pain
Keywords: upper back/neck/shoulder muscle spasm
MeSH Terms: conditions — Back Pain | interventions — Guaifenesin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): Guaifenesin 1 tablet BID
  Interventions: Drug: Guaifenesin
- Arm 2 (Experimental): Guaifenesin 2 tablets BID
  Interventions: Drug: Guaifenesin
- Arm 3 (Placebo Comparator): Placebo 1 tablet BID
  Interventions: Drug: Placebo
- Arm 4 (Placebo Comparator): Placebo 2 tablets BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guaifenesin — high and low dose of Guaifenesin each given twice daily over a 4-day treatment period
  Arms: Arm 1; Arm 2
Drug: Placebo — no active ingredient
  Arms: Arm 3; Arm 4

SUMMARY:
Explore the clinical efficacy of 7-day treatment regimens of guaifenesin in order to investigate the evidence that guaifenesin is an effective treatment for upper back/neck/shoulder muscle spasm/stiffness and pain.

ELIGIBILITY:
Inclusion Criteria:

* Paticipant presents with a new episode of acute upper back/neck/shoulder pain and muscle spasm that:

  1. is at least 30 days from previous episode.
  2. has an onset occurred within 48 hours of Visit 1.
  3. has symptoms consistent with a clinical diagnosis as per the physical examination at Visit 1.
  4. has a subject-rated muscle spasm score and a pain score of at least 40 out of 100 on a 100mm VAS.
* Paticipant has a normal neurological examination.

Exclusion Criteria:

* Medical history: a) Paticipant has a known or suspected intolerance or hypersensitivity to guaifenesin or methocarbamol (or closely related compounds) or any of their stated ingredients. b) Paticipant has history of upper back pain with active hypersensitive spots - trigger point in the muscles of upper back/neck/shoulder/maxillofacial regions. c) Paticipant has a current or recent history of liver and/or kidney disease, neck/back/shoulder injuries, spinal disc disease, myocardial infarction (<12 months from Visit 1) and osteoporosis. d) Subjects have history of other chronic pain e.g. headache, osteoarthritis, arthritis, lower back pain etc.
* Medications: a) Paticipant has used a muscle relaxant or narcotic within 2 weeks of Visit 1. b) Paticipant has used monoamine oxidase inhibitors or selegiline within 2 weeks of Visit 1 c) Currently using tricyclic antidepressants, lithium, anticoagulants, or tramadol.
* Paticipant is involved in a workers compensation case.
* Paticipant is unlikely to refrain from using analgesics, NSAIDs, and other muscle relaxants for the duration of the study, with the exception of cardioprotective doses of aspirin (i.e., ≤ 325 mg/day).
* Paticipant is unlikely to refrain from physical therapy, massage therapy, acupuncture, heat treatment, spas, etc for the duration of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (5):
  - Med Investigations, Fair Oaks, California
  - San Diego Sports Medicine and Family Health Center, San Diego, California
  - Radiant Research - Cincinnati, Cincinnati, Ohio
  - Radiant Research, Inc. - TX, San Antonio, Texas
  - J. Lewis Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at multiple clinical sites
Pre-assignment Details: Male or female participants aged 18-65 years (inclusive) with acute onset upper back/neck/shoulder muscle spasm and pain were recruited in this study
Groups:
- Guaifenesin 600mg: Guaifenesin 600mg Extended Release Tablet taken orally with 150ml of water twice daily (BID), for 7 consecutive days
- Placebo Matching Guaifenesin 600mg: 1 placebo tablet matching Guaifenesin 600mg Extended Release Tablet taken orally with 150ml of water BID, for 7 consecutive days
- Guaifenesin 1200mg: 2 Guaifenesin 600mg Extended Release Tablets taken orally with 150ml of water BID, for 7 consecutive days
- Placebo Matching Guaifenesin 1200mg: 2 placebo tablets matching Guaifenesin 1200mg Extended Release Tablets taken orally with 150ml of water BID, for 7 consecutive days
Period: Overall Study
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Started | 25 | 15 | 25 | 14
Completed | 25 | 15 | 24 | 14
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg | Total
Number analyzed (Participants) | 25 | 15 | 24 | 14 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.2 (11.87) | 43.8 (10.35) | 45.3 (10.62) | 47.3 (13.92) | 45.9 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 12 | 6 | 35
  Male | 17 | 6 | 12 | 8 | 43

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline of Both AM and PM Spasm Assessment Scores
Description: The score was measured as 'assessment at baseline' minus 'assessment after treatment' over 7 day period (mean of all AM and PM changes from baseline). Measurements were based on an 11 categorical Numerical Rating Scale (NRS) with a range from 0 - no spasm to 10 - unbearable spasm.
Time Frame: 7 Days
Population: Efficacy analysis was conducted on the intention-to-treat (ITT) population, defined as all subjects who received at least one dose of study medication and who had at least one post-baseline efficacy assessment. Subjects were analyzed according to the treatment to which they were randomized.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Placebo Matching Guaifenesin 600mg: 1 placebo tablet matching Guaifenesin 600mg Extended Release Tablet taken orally with 150ml of water BID for 7 consecutive days
- Placebo Matching Guaifenesin 1200mg: 2 placebo tablets matching Guaifenesin 1200mg Extended Release Tablets taken orally with 150ml of water BID for 7 consecutive days
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Number analyzed (Participants) | 25 | 15 | 24 | 13
Score on a Scale | 1.66 (1.806) | 1.87 (1.644) | 1.91 (1.541) | 1.54 (1.203)
Statistical Analysis 1: Comparison: Guaifenesin 600mg vs Placebo Matching Guaifenesin 600mg; Null hypotheses was tested as: H01: There was no difference in the mean change from baseline of muscle spasm score between Guaifenesin 600mg and placebo. H02: There was no difference in the mean change from baseline of muscle spasm score between Guaifenesin 1200mg and placebo. H03: There was no difference in the mean change from baseline of muscle spasm score between Guaifenesin 1200mg and Guaifenesin 600mg; Test type: Superiority or Other; p = 0.68, t-test, 2 sided — P-value was associated with t-test for difference of LS means; The model included factors for treatment (as a fixed effect) and site (as a random effect); Least Squares Means Difference = -0.21, 95% CI 2-sided [-1.23 to 0.80] — Least Square mean from Mixed Model including factors for treatment (as a fixed effect) and site (as a random effect). Difference was First named treatment - second named treatment
Statistical Analysis 2: Comparison: Guaifenesin 1200mg vs Placebo Matching Guaifenesin 1200mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.52, t-test, 2 sided — P-value associated with t-test for difference of LS means; Least Squares Means Difference = 0.35, 95% CI 2-sided [-0.72 to 1.42] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Guaifenesin 600mg vs Guaifenesin 1200mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.58, t-test, 2 sided — P-value associated with t-test for difference of LS means; Least Squares Means Difference = 0.24, 95% CI 2-sided [-0.64 to 1.13] — Least Square mean from Mixed Model including factors for treatment (as a fixed effect) and site (as a random effect). Difference was Second named treatment - first named treatment

2. Secondary Outcome: Mean Change From Baseline of Both AM and PM NRS Muscle Stiffness Assessment Scores
Description: The score was measured as 'assessment at baseline' minus 'assessment after treatment' over 7 day period (mean of all AM and PM changes from baseline). Measurements were based on an 11 categorical Numerical Rating Scale (NRS) with a range from 0 - no stiffness to 10 - unbearable stiffness.
Time Frame: 7 Days
Population: Efficacy analysis were conducted on the intention-to-treat (ITT) population, defined as all subjects who receive at least one dose of study medication and who had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Number analyzed (Participants) | 25 | 15 | 24 | 13
Score on a scale | 1.90 (1.684) | 2.09 (1.225) | 1.87 (1.630) | 1.77 (1.214)

3. Secondary Outcome: Mean Change From Baseline of Both AM and PM NRS Tension Assessment Scores
Description: The score was measured as 'assessment at baseline' minus 'assessment after treatment' over 7 day period (mean of all AM and PM changes from baseline). Measurements were based on an 11 categorical Numerical Rating Scale (NRS) with a range from 0 - no tension to 10 - unbearable tension.
Time Frame: 7 Days
Population: Efficacy analysis were conducted on the intention-to-treat (ITT) population, defined as all subjects who received at least one dose of study medication and who had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Number analyzed (Participants) | 25 | 15 | 24 | 13
Score on a scale | 1.74 (1.721) | 1.98 (1.496) | 1.97 (1.540) | 1.54 (1.678)

4. Secondary Outcome: Mean Change From Baseline of Both AM and PM NRS Pain Assessment Scores
Description: The score was measured as 'assessment at baseline' minus 'assessment after treatment' over 7 day period (mean of all AM and PM changes from baseline). Measurements were based on an 11 categorical Numerical Rating Scale (NRS) with a range from 0 - no pain to 10 - unbearable pain.
Time Frame: 7 Days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Number analyzed (Participants) | 25 | 15 | 24 | 13
Score on a scale | 1.65 (2.028) | 2.41 (1.376) | 2.14 (1.539) | 1.41 (0.995)

5. Secondary Outcome: Mean Change From Baseline of Both AM and PM NRS Discomfort Assessment Scores
Description: The score was measured as 'assessment at baseline' minus 'assessment after treatment' over 7 day period (mean of all AM and PM changes from baseline). Measurements were based on an 11 categorical Numerical Rating Scale (NRS) with a range from 0 - no discomfort to 10 - unbearable discomfort.
Time Frame: 7 Days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Number analyzed (Participants) | 25 | 15 | 24 | 13
Score on a scale | 1.95 (1.824) | 2.57 (1.406) | 2.33 (1.668) | 1.12 (1.459)

6. Secondary Outcome: Muscle Relaxation Scores
Description: The score was measured as mean of both AM and PM assessment scores at Days 4 and 7. Measurements were based on a 5 categorical scale: 0 - no relaxation, 1- a little relaxation, 2 - fair relaxation, 3 - good relaxation, 4 - complete muscle relaxation.
Time Frame: 4 Days, 7 Days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Number analyzed (Participants) | 25 | 15 | 24 | 13
Score on a scale
  Degree of Muscle Relaxation at Day 4 | 1.80 (0.829) | 1.90 (0.507) | 1.85 (0.759) | 1.35 (0.826)
  Degree of Muscle Relaxation at Day 7 | 1.86 (0.860) | 2.27 (0.980) | 2.17 (1.007) | 1.69 (1.146)

7. Secondary Outcome: Upper Back/Neck/Shoulder Pain Disability (Vernon-Mior) Index Scores
Description: Vernon-Mior upper back/neck/shoulder components were assessed before the treatment and at Days 4 and 7. Each component (pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation) was assessed based on a 6-point categorical scale (1 to 6), with 1 being the most positive and 6 being the worst.
Time Frame: Before treatment, 4 Days, 7 Days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Number analyzed (Participants) | 25 | 15 | 24 | 13
Score on a scale
  Pain Intensity-before treatment | 3.88 (0.781) | 3.67 (0.816) | 3.25 (0.897) | 3.62 (0.650)
  Pain Intensity-Day 4 | 2.72 (0.980) | 2.53 (0.834) | 2.29 (0.955) | 2.83 (0.577)
  Pain Intensity-Day 7 | 2.48 (0.918) | 2.20 (0.862) | 1.88 (0.797) | 1.92 (0.641)
  Personal Care-before treatment | 1.96 (0.735) | 2.07 (0.799) | 2.00 (0.780) | 2.00 (0.816)
  Personal Care-Day 4 | 1.72 (0.678) | 1.60 (0.632) | 1.50 (0.511) | 1.75 (0.754)
  Personal Care-Day 7 | 1.60 (0.707) | 1.33 (0.488) | 1.29 (0.550) | 1.46 (0.519)
  Lifting-before treatment | 3.04 (1.060) | 3.13 (1.302) | 2.92 (1.139) | 3.15 (1.144)
  Lifting-Day 4 | 2.80 (1.258) | 2.27 (1.100) | 2.58 (1.139) | 2.42 (1.311)
  Lifting-Day 7 | 2.56 (1.387) | 2.00 (1.309) | 2.04 (0.999) | 2.00 (1.291)
  Reading-before treatment | 3.00 (1.225) | 2.67 (0.976) | 2.29 (1.042) | 2.92 (1.038)
  Reading-Day 4 | 2.40 (0.913) | 2.20 (1.014) | 1.88 (0.947) | 2.38 (0.650)
  Reading-Day 7 | 2.00 (0.707) | 1.73 (0.799) | 1.58 (0.776) | 1.85 (0.689)
  Headache-before treatment | 1.72 (0.980) | 1.87 (0.743) | 1.79 (0.932) | 2.23 (0.832)
  Headache-Day 4 | 1.76 (1.165) | 1.67 (0.900) | 2.04 (1.367) | 2.23 (0.832)
  Headache-Day 7 | 1.60 (0.913) | 1.67 (0.617) | 1.75 (1.152) | 2.00 (0.816)
  Concentration-before treatment | 2.12 (1.013) | 2.20 (1.320) | 1.88 (0.992) | 2.08 (0.494)
  Concentration-Day 4 | 1.75 (0.737) | 1.60 (0.507) | 1.54 (0.588) | 2.00 (0.707)
  Concentration-Day 7 | 1.76 (0.831) | 1.53 (0.640) | 1.46 (0.588) | 1.62 (0.506)
  Work-before treatment | 2.64 (1.186) | 2.80 (1.014) | 2.50 (0.834) | 3.00 (1.354)
  Work-Day 4 | 2.20 (0.957) | 2.13 (0.915) | 1.92 (0.929) | 2.46 (0.877)
  Work-Day 7 | 1.96 (0.841) | 1.73 (0.799) | 1.75 (0.847) | 2.08 (1.382)
  Driving-before treatment | 3.12 (1.424) | 2.67 (0.816) | 2.21 (0.779) | 3.00 (1.225)
  Driving-Day 4 | 2.56 (1.530) | 2.13 (1.302) | 1.79 (0.779) | 2.38 (1.193)
  Driving-Day 7 | 2.48 (1.503) | 2.00 (1.254) | 1.46 (0.509) | 2.15 (1.345)
  Sleeping-before treatment | 3.16 (1.179) | 3.47 (1.356) | 2.96 (1.083) | 3.23 (1.363)
  Sleeping-Day 4 | 2.76 (1.363) | 2.67 (1.291) | 2.42 (1.139) | 2.92 (1.188)
  Sleeping-Day 7 | 2.56 (1.193) | 2.20 (0.862) | 2.04 (1.083) | 1.92 (0.954)
  Recreation-before treatment | 3.44 (1.261) | 3.27 (1.100) | 2.88 (0.992) | 3.23 (1.235)
  Recreation-Day 4 | 2.44 (1.121) | 2.40 (1.121) | 2.17 (0.917) | 2.54 (1.266)
  Recreation-Day 7 | 2.29 (1.083) | 1.73 (0.594) | 1.88 (1.035) | 2.08 (1.320)

8. Secondary Outcome: Global Assessment of Treatment Helpfulness (GATH)
Description: Measured as an overall qualitative score on a 5 point categorical scale: 0-poor, 1-fair, 2-good, 3-very good and 4-excellent.
Time Frame: 4 Days, 7 Days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Number analyzed (Participants) | 25 | 15 | 24 | 13
Score on a scale
  Global Assessment of Treatment Helpfulness- Day 4 | 1.48 (1.194) | 1.53 (0.743) | 1.63 (0.824) | 0.85 (0.899)
  Global Assessment of Treatment Helpfulness- Day 7 | 1.56 (1.083) | 1.73 (1.163) | 1.71 (0.999) | 1.38 (1.121)

9. Secondary Outcome: Global Assessment of Sleep Disturbance (GASD)
Description: Categorized after treatment as: 'decreased', 'increased' or 'stayed the same'.
Time Frame: 7 Days
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Number analyzed (Participants) | 25 | 15 | 24 | 13
participants
  Global Assessment of Sleep Disturbance-Decreased | 8 | 8 | 10 | 7
  Global Assessment of Sleep Disturbance-Increased | 1 | 0 | 2 | 1
  Global Assessment of Sleep Disturbance-Stayed same | 16 | 7 | 12 | 5

10. Secondary Outcome: Global Assessment of Headache Frequency (GAHF)
Description: Categorized after treatment as: 'decreased', 'increased' or 'stayed the same'.
Time Frame: 7 Days
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Number analyzed (Participants) | 25 | 15 | 24 | 13
participants
  Headache frequency-decreased | 9 | 9 | 7 | 4
  Headache frequency-increased | 3 | 0 | 1 | 0
  Headache frequency-stayed same | 13 | 6 | 16 | 9

11. Secondary Outcome: Global Assessment of Headache Intensity (GAHI)
Description: Categorized after treatment as: 'decreased', 'increased' or 'stayed the same'.
Time Frame: 7 Days
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Number analyzed (Participants) | 25 | 15 | 24 | 13
participants
  Headache Intensity-decreased | 10 | 9 | 9 | 4
  Headache Intensity-increased | 1 | 0 | 1 | 0
  Headache Intensity-stayed same | 14 | 6 | 14 | 9

ADVERSE EVENTS:
Time Frame: All adverse events were collected from the start of the investigational product, and until 7 days following last administration of the investigational product.
Arm/Group | Guaifenesin 600mg | Placebo Matching Guaifenesin 600mg | Guaifenesin 1200mg | Placebo Matching Guaifenesin 1200mg
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/15 | 0/24 | 0/14
Other Adverse Events (participants affected / at risk) | 7/25 | 1/15 | 6/24 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guaifenesin 600mg (N=25) | Placebo Matching Guaifenesin 600mg (N=15) | Guaifenesin 1200mg (N=24) | Placebo Matching Guaifenesin 1200mg (N=14)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.